CLINICAL TRIAL: NCT02931279
Title: Evaluation of the Efficacy and Safety of the Cervical Posterior Fixation System PASS OCT®
Brief Title: PASS OCT® Post-market Clinical Follow-up
Status: Completed | Type: Observational
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: 1701
Record Dates: First submitted 2016-06-27; First posted 2016-10-13 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Intervertebral Disc Disease; Spondylolisthesis; Spinal Stenosis; Spinal Neoplasms; Spinal Fractures
MeSH Terms: conditions — Intervertebral disc disease; Spondylolisthesis; Spinal Stenosis; Spinal Neoplasms; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PASS OCT® Spinal System — Posterior osteosynthesis of the cervical and upper thoracic spine

SUMMARY:
Prospective, multicenter non comparative and observational study (post-market clinical follow-up).

Patients operated with PASS OCT® manufactured by MEDICREA® INTERNATIONAL between July 2016 and July 2017.

The inclusion period will be 12 months and the follow-up 24 months

DETAILED DESCRIPTION:
The primary endpoint is to evaluate the safety of the PASS OCT® system.

The secondary endpoints are to analyze the efficacy of the system with several point of view:

* The quality of fusion and the time of fusion through X rays
* the pain with VAS
* the quality of life thanks to questionnaires: NDI (Neck Disability Index) and JOA for myelopathy
* the daily of the patient: return to work, sport
* the surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient with

  * degenerative disc disease or,
  * spondylolisthesis, or
  * spinal stenosis, or
  * trauma, or
  * atlanto-axial fractures with instability or
  * cervical tumors.
* Patient operated with PASS OCT®
* Patient > 18 years
* Patient affiliated to health care insurance (social security in France)
* Patient able to complete a self-administered questionnaire
* Patient able to understand the protocol and the planning visit
* Patient able to sign an informed consent form

Exclusion Criteria:

* Patient unable or unwilling to sign an informed consent form
* Patient unable to complete a self-administered questionnaire
* Pregnant patient or intending to get pregnant within the next 3 years
* Patient judged as non-compliant by the investigator or not able to come back for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who need immobilization and stabilization of spinal segments as an adjunct to fusion of the occipital, cervical and/or upper thoracic spine (Occiput-T3).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 months postoperatively
  To quantify and describe adverse events

SECONDARY OUTCOMES:
Fusion | 1-6 months, 12 months, 24 months postoperatively
  Radiological assessment of bony fusion
Disability | 1-6 months, 12 months, 24 months postoperatively
  To assess disability using NDI score
Quality of life | 1-6 months, 12 months, 24 months postoperatively
  To assess quality of life through mJOA scoring system
Pain | 1-6 months, 12 months, 24 months postoperatively
  To assess pain using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Fuentes, MD, Principal Investigator — Hopital la Timone, Marseille
Locations (1):
- Hopital la Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: No